CLINICAL TRIAL: NCT00337207
Title: A Phase II Safety Study of Bevacizumab in Patients With Multiple Recurrent or Progressive Malignant Gliomas
Brief Title: Bevacizumab in Treating Patients With Recurrent or Progressive Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Raizer, Jeffrey Raizer, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 05C3; NU-05C3 (Other: Northwestern University Cancer Center); STU00005237 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult gliosarcoma; recurrent adult brain tumor; adult anaplastic astrocytoma; adult giant cell glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms; Astrocytoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin (Experimental)
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — Bevacizumab 15 mg/kg every 3 weeks over 30 to 90 minutes. One cycle = 3 weeks. Treatment continues until progressive disease or unacceptable toxicity.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well bevacizumab works in treating patients with recurrent or progressive glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of single-agent bevacizumab in the treatment of patients with recurrent or progressive malignant glioma.
* Determine the efficacy of bevacizumab, in terms of progression-free survival at 6 months, in these patients.
* Assess changes in tumoral blood flow based on magnetic resonance (MR) perfusion and tissue changes by MR spectroscopy.

OUTLINE: This is a pilot study.

Patients receive bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma, including the following:

  * Glioblastoma multiforme
  * Gliosarcoma
  * Anaplastic astrocytoma or anaplastic glioma
  * Malignant glioma not otherwise specified
* Evidence of tumor recurrence or progression by MRI or CT scan with contrast

  * CT scan or MRI must be performed ≤ 96 hours post-operatively (≤ 2 weeks prior to study registration) or 4-6 weeks post-operatively to assess residual disease in patients who have undergone recent resection of recurrent or progressive tumor

    * Steroid dosage must have been stable for ≥ 5 days
* Failed ≥ 1 prior systemic treatment with chemotherapy or biologic agents (excluding polifeprosan 20 with carmustine implant [Gliadel wafers])
* Failed prior external-beam radiotherapy
* If received prior interstitial brachytherapy or stereotactic radiosurgery, true progressive disease (rather than radiation necrosis) must be confirmed by positron emission tomography, single-photon emission computer tomography with thallium, magnetic resonance (MR) spectroscopy, MR perfusion, or surgical documentation

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy > 8 weeks
* WBC > 3,000/mm³
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 10 g/dL (transfusion allowed)
* SGOT and SGPT < 1.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Creatinine < 1.5 mg/dL
* Blood pressure ≤ 150/100 mm Hg
* No unstable angina
* No New York Heart Association class II-IV congestive heart failure
* No stroke or myocardial infarction within the past 6 months
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* Urine protein:creatinine ratio < 1.0
* No significant medical illness that would preclude study participation or cannot be adequately controlled with appropriate therapy
* No other serious medical illness or infection
* No disease that would obscure toxicity or dangerously alter drug metabolism
* No significant traumatic injury within the past 28 days
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious, nonhealing wound, ulcer, or bone fracture
* No history of any other cancer (except nonmelanoma skin cancer or carcinoma in situ of the cervix) unless cancer is in complete remission and patient is off all therapy for that cancer for ≥ 3 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior surgery for recurrent or progressive disease and recovered
* More than 28 days since prior major surgical procedure or open biopsy
* At least 4 weeks since prior cytotoxic therapy (6 weeks for nitrosoureas)
* At least 2 weeks since prior vincristine
* At least 3 weeks since prior procarbazine hydrochloride
* At least 1 week since prior noncytotoxic agents (e.g., interferon, tamoxifen, thalidomide, or isotretinoin)

  * Radiosensitizer does not count
* At least 4 weeks since prior experimental biologic agents (e.g., epidermal growth factor receptor [EGFR] inhibitors)
* More than 7 days since prior minor surgery, such as fine-needle aspirations or core biopsies
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No concurrent enzyme-inducing anticonvulsants (EIACs)

  * Patients on EIACs must switch to nonenzyme-inducing convulsants ≥ 2 weeks prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Raizer, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois

REFERENCES:
- [Result] Raizer JJ, Gallot L, Cohn R, et al.: A phase II safety study of bevacizumab in patients with multiple recurrent or progressive malignant gliomas. [Abstract] J Clin Oncol 25 (Suppl 18): A-2079, 94s, 2007.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Neuro-Oncology outpatient clinic and inpatient services between the dates of March 16, 2006 and June 5, 2008.
Groups:
- Study Treatment: All patients received bevacizumab 15 mg/kg every 3 weeks until progressive disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | Study Treatment
Started | 55
Completed | 52
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.91 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 47
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55
Diagnosis [Number; unit: Participants] — Patients with histologically proven malignant gliomas were eligible to be enrolled including the following diagnoses: glioblastoma multiforme (GBM), gliosarcoma, anaplastic astrocytoma (AA), anaplastic oligodendronglioma, anaplastic mixed glioma or malignant glioma NOS (not otherwise specified).
  Participants
    Glioblastoma multiforme (GBM) | 44
    Anaplastic astrocytoma (AA) | 7
    Gliosarcoma | 0
    Anaplastic oligodendronglioma | 4
    Anaplastic mixed glioma | 0
    Malignant glioma NOS (not otherwise specified) | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety of Treatment
Description: Safety of treatment will be defined by the number of patients that experience grade 3 and 4 adverse events where causal relationship with bevacizumab cannot be completely ruled out. Adverse events will be graded using Common Terminology Criteria for Adverse Events v3.0 (CTCAE) where:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: From treatment initiation, throughout treatment and up to 30 days post-treatment, for up to 1 year.
Population: All patients that receive at least one dose of study treatment are evaluable for toxicity
Measure: Number; unit: participants
Groups:
- Bevacizumab Treatment: All patients received bevacizumab 15 mg/kg every 3 weeks until progressive disease or unacceptable toxicity.
Arm/Group | Bevacizumab Treatment
Number analyzed (Participants) | 55
participants
  Bowel perforation | 1
  DVT | 1
  Fatigue | 5
  Headache | 1
  Lack of drive | 1
  Rectal bleeding | 2

2. Primary Outcome: Progression-free Survival at 6 Months
Description: The number of patients experiencing progression free survival (PFS) was calculated at the 6-month time point.
Time Frame: After all patients have surpassed the 6 month post-treatment timepoint
Population: 1 patient became deceased due to toxicity prior to the 6 month time point and thus, was not evaluable for the 6 month progression free survival endpoint.
Measure: Number; unit: Participants
Arm/Group | Study Treatment
Number analyzed (Participants) | 54
Participants
  # of Patients Experiencing PFS at 6 months | 13
  # of Patients Who Progressed Prior to 6 months | 41

3. Primary Outcome: Tumoral Blood Flow Changes
Description: To assess changes in tumoral blood flow based on MR Perfusion and tissue changes by MR spectroscopy.
Time Frame: Before and after treatment
Population: This was an optional outcome measure. Data was not collected or analyzed for this outcome measure.
Arm/Group | Bevacizumab Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From time of first study treatment up to 30 days after the last dose (total time frame was variable by patient).
Description: All patients were evaluable for toxicity from the time of their first treatment with bevacizumab. Patients continued on treatment until disease progression or unacceptable toxicity, thus the evaluation period was different for each patient.
Arm/Group | Study Treatment
Serious Adverse Events (participants affected / at risk) | 9/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment (N=55)
Hemorrhage - GI (rectal) (Gastrointestinal disorders) | 1 (1)
Perforation - GI (bowel) (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Thrombosis/embolism (venous) (Vascular disorders) | 1 (1)
Death due to disease progression (General disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment (N=55)
Fatigue (General disorders) | 27 (27)
Hemorrhage (Vascular disorders) | 15 (15)
Hypertension (Cardiac disorders) | 12 (12)
Pain - headache (General disorders) | 10 (10)
Infection (Infections and infestations) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 11 (11)
Memory impairment (Nervous system disorders) | 7 (7)
Neuropathy - motor (Nervous system disorders) | 3 (3)
Neuropathy - sensory (Nervous system disorders) | 3 (3)
Personality/behavioral (Psychiatric disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4)
Elevated transaminases - AST/ALT (Metabolism and nutrition disorders) | 9 (9)
Weight loss (General disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pain - arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain - Not otherwise specified (General disorders) | 3 (3)
Renal - Other (hematuria) (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes